CLINICAL TRIAL: NCT01327872
Title: A Randomized, Open-Label, 4-Group, 2-Period Replicate Design Study to Evaluate Within- and Between-Subject Variability in Exposure of Two Lots of E5501 20 mg Tablets, Administered as Single Doses of 40 mg, in the Fasted and Fed Conditions to Healthy Subjects
Brief Title: Subject Variability in Two Lots of E5501 Administered to Fed and Fasted Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E5501-G000-010
Record Dates: First submitted 2011-03-30; First posted 2011-04-04 (Estimated); Last update posted 2012-03-09 (Estimated); Status verified 2012-03

CONDITIONS: Purpura, Thrombocytopenic, Idiopathic; Acute Idiopathic Thrombocytopenic Purpura; Chronic Thrombocytopenia
Keywords: Idiopathic Thrombocytopenia Purpura(ITP); Acute and Chronic Thrombocytopenia Associated with Chronic Liver Disease; TLD
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A (Experimental)
  Interventions: Drug: E5501 40 mg 2 x 20-mg tablets, orally, fasted
- Treatment B (Experimental)
  Interventions: Drug: E5501 40 mg 2 x 20-mg tablets, orally, with food
- Treatment C (Experimental)
  Interventions: Drug: E5501 40mg 2 x 20-mg tablets, orally, fasted
- Treatment D (Experimental)
  Interventions: Drug: E5501 40 mg 2 x 20-mg tablets, orally, with food

INTERVENTIONS:
Drug: E5501 40 mg 2 x 20-mg tablets, orally, fasted — single 40 mg dose (2 x 20-mg tablets) of Lot P01008ZZA in the fasted condition
  Arms: Treatment A
Drug: E5501 40 mg 2 x 20-mg tablets, orally, with food — single 40 mg dose (2 x 20-mg tablets) of Lot P01008ZZA in the fed condition
  Arms: Treatment B
Drug: E5501 40mg 2 x 20-mg tablets, orally, fasted — single 40 mg dose (2 x 20-mg tablets) of Lot P01009ZZA in the fasted condition
  Arms: Treatment C
Drug: E5501 40 mg 2 x 20-mg tablets, orally, with food — single 40 mg dose (2 x 20-mg tablets) of Lot P01009ZZA in the fed condition
  Arms: Treatment D

SUMMARY:
This will be a randomized, open-label, four-group, two-period, replicate design study to evaluate the effect of food on within and between subject variability in second generation formulation 20-mg tablet strengths, Lots P01008ZZA and P01009ZZA, administered as single doses of 40mg to 84 healthy male and female subjects. The study is powered to detect both a reduction in either the within or between subject variability (coefficient of variation [CV]%) of approximately 35%.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, double-blind, randomized, placebo-controlled, dose-ranging, parallel-group study. The PK and PK/PD relationship of AKR-501 will also be studied. Approximately 65 eligible patients will be randomized in a 3:3:3:3:1 ratio in a double-blinded fashion into one of five parallel treatment groups to receive daily doses of either AKR-501 2.5, 5, 10 or 20 mg or placebo for 28 days, respectively. Each AKR-501 dosing group will consist of 15 patients while the placebo group will consist of 5 patients. All study patients will be evaluated weekly (Days 3, 5, 7, 14, 21 and 28) for safety, efficacy, and (Days 7, 14, 21, and 28) AKR-501 pharmacokinetics while receiving study treatment with a final assessment for safety and effectiveness to be done 2 weeks after the last study dose (Day 42).

ELIGIBILITY:
Inclusion criteria:

* Normal healthy male or female subjects age greater than or equal to 18 years and less than or equal to 55 years
* Body mass index greater than or equal to 18 and less than or equal to 32kg/m2 at Screening
* Platelet count greater than or equal to 120x109/L and less than or equal to 250x109/L
* Women of childbearing potential must agree to use a highly effective method of contraception, other than estrogen-based hormonal contraceptives, during the Randomization Phase of the study

Exclusion Criteria:

* Evidence of clinically significant cardiovascular, hepatic, gastrointestinal, renal, respiratory, endocrine, hematologic, neurologic, or psychiatric disease or abnormalities or a known history of any gastrointestinal surgery that could impact PK of the study drug
* Agents associated with thrombotic events (including oral contraceptives) must be discontinued within 30 days of first study drug administration
* Evidence of organ dysfunction or any clinically significant deviation from normal in their medical history, e.g., history of splenectomy
* History of venous or arterial thrombotic disease or other hypercoaguable state
* Hemoglobin less than lower limit of normal (LLN) levels (females 7.1 mmol/L, males 8.1 mmol/L

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2011-02; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time course profile (AUC) and maximum observed plasma concentration (Cmax) under fasted and fed conditions | 8 weeks

SECONDARY OUTCOMES:
To evaluate the comparison of the overall effect of food on the bioavailability of E5501 relative to the fasted condition as measured by AUC(0-inf) and Cmax | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Johnson, Study Director — Eisai Inc.
Locations (1):
- PRA Early Development Services, Zuidlaren, Netherlands